CLINICAL TRIAL: NCT00394199
Title: A Randomized, Double-blind, Active-controlled, Parallel Group, Stratified, Multi-center, 12-week Study Comparing the Safety & Efficacy of Fluticasone and Formoterol Combination (FlutiForm(tm) 100/10 µg Twice Daily) in a Single Inhaler (SkyePharma HFA pMDI) With the Administration of Fluticasone (100 µg Twice Daily) and Formoterol (10 µg Twice Daily) Alone in Adolescent & Adult Patients With Mild to Moderate Asthma
Brief Title: Comparison of New Combination Inhaler (FlutiForm HFA MDI 100/10 µg) Versus Fluticasone & Formoterol Administered Alone in Patients With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SkyePharma AG (Industry)
Responsible Party: SkyePharma AG, SkyePharma AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SKY2028-3-002
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Asthma
Keywords: Asthma; Fluticasone Propionate; formoterol fumarate; Pressurized metered dose inhaler; Hydrofluoroalkane; Mild to Moderate Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 1 (Experimental): FlutiForm 100/10ug
  Interventions: Drug: Fluticasone propionate/Formoterol Fumarate 100/10
- 2 (Experimental): Fluticasone 100
  Interventions: Drug: Fluticasone propionate 100
- 3 (Active Comparator): Formoterol 10
  Interventions: Drug: Formoterol fumarate 10

INTERVENTIONS:
Drug: Fluticasone propionate/Formoterol Fumarate 100/10 — FlutiForm 100/10ug is a HFA pMDI that delivers 50ug of Fluticasone propionate per actuation and 5ug of Formoterol fumarate per actuation. Patients will take 2 actuations BID for 12 weeks.
  Other Names: Flutiform 100/10
  Arms: 1
Drug: Fluticasone propionate 100 — Fluticasone 100 is a HFA pMDI that delivers 50ug of Fluticasone propionate per actuation. Patients will take 2 actuations BID for 12 weeks.
  Other Names: Fluticasone 100
  Arms: 2
Drug: Formoterol fumarate 10 — Formoterol 10ug is a HFA pMDI that delivers 5ug of Formoterol fumarate per actuation. Patients will take 2 actuations BID for 12 weeks.
  Other Names: SKP Formoterol 10
  Arms: 3

SUMMARY:
To compare the efficacy and safety of the fixed combination asthma drug Flutiform HFA MDI with its two components administered alone, fluticasone propionate and formoterol fumarate, in adult and adolescent patients with mild to moderate asthma.

ELIGIBILITY:
* Ages eligible for study: 12 years and above
* Genders eligible for study: both
* Prior steroid use: steroid-requiring or steroid-free

Inclusion Criteria:

* History of asthma for at least 12 months
* For steriod-requiring patients, documented use of inhaled corticosteroid for at least 4 weeks prior to Screening Visit
* For steroid-free patients, no history of inhaled steroid asthma medication for at least 12 weeks prior to Screening Visit
* Demonstrate FEV-1 of 60-85% of predicted normal values at Screening and Baseline Visit
* Documented reversibility of 15% within 12 months of Screening or at Screening Visit (15% increase from pre-FEV-1 levels following albuterol inhalation or nebulized albuterol administration)
* Symptoms of asthma during Run-in
* Females of childbearing potential must have a negative urine pregnancy test at Screening and Baseline Visits. Females are eligible only if they are not pregnant or lactating, and are either sterile, or using acceptable methods of contraception.
* Must otherwise be healthy
* Provide written informed consent. Wishes of minors must be respected.

Exclusion Criteria:

Patients will not be eligible for the study if they meet any of the following criteria:

* Life-threatening asthma within the past year or during the Run-In Period.
* History of systemic corticosteroid medication within 3 months before the Screening Visit.
* History of omalizumab use within past 6 months.
* History of leukotriene receptor antagonist use, e.g., montelukast, within past week.
* Current evidence or history of any clinically significant disease or abnormality including uncontrolled hypertension, uncontrolled coronary artery disease, congestive heart failure, myocardial infarction, or cardiac dysrhythmia.
* Upper or lower respiratory infection within 4 weeks prior to Screening Visit or during Run-In Period.
* Significant, non-reversible, pulmonary disease (e.g., chronic obstructive pulmonary disease [COPD], cystic fibrosis, bronchiectasis).
* Known Human Immunodeficiency Virus (HIV)-positive status.
* Smoking history equivalent to "10 pack years".
* Current smoking history within 12 months prior to Screening Visit.
* Current evidence or history of alcohol and/or substance abuse within 12 months prior to Screening Visit.
* Patients who are confined in institution.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2006-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change in Forced Expiratory volume in 1 s (FEV-1) from morning predose at Baseline (Week 0) to predose at Week 12 | Week 0 and 12

SECONDARY OUTCOMES:
Other pulmonary function tests including forced vital capacity (FVC) and peak expiratory flow rate (PEFR). | Whole duration of study
Clinical endpoints (frequency of asthma exacerbations and patient data captured in diary including daily morning and evening PEFR). | Whole duration of study
Safety variables include adverse events, ECGs, clinical laboratory tests and vital signs. | Whole duration of study

CONTACTS AND LOCATIONS:
Locations (41):
- United States (29):
  - Research Site, Birmingham, Alabama
  - Research Site, Mission Viejo, California
  - Research Site, Orange, California
  - Research Site, San Jose, California
  - Research Site, Vista, California
  - Research Site, Denver, Colorado
  - Research Site, Lilburn, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Park City, Kansas
  - Research Site, Bethesda, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Center, Stevensville, Michigan
  - Research Site, Elizabeth, New Jersey
  - Research Center, Rochester, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Sylvania, Ohio
  - Research Site, Easton, Pennsylvania
  - Research Site, Lincoln, Rhode Island
  - Research Site, Greenville, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Katy, Texas
  - Research Site, New Braunfels, Texas
  - Research Site, Waco, Texas
  - Research Site, South Burlington, Vermont
  - Research Site, Greenfield, Wisconsin
- Canada (12):
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Center, London, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saint Foy, Quebec
  - Research Site, Trois-Rivières, Quebec

REFERENCES:
- [Derived] Pearlman DS, LaForce CF, Kaiser K. Fluticasone/Formoterol combination therapy compared with monotherapy in adolescent and adult patients with mild to moderate asthma. Clin Ther. 2013 Jul;35(7):950-66. doi: 10.1016/j.clinthera.2013.05.012. PMID 23870606